CLINICAL TRIAL: NCT02455323
Title: Influence of Spinal Manipulation and Suboccipipital Inhibition as a Complementary Therapy for Tension Headache in Quality of Life: A Randomized Controlled Trial
Brief Title: The Influence of Manual Therapy in the Quality of Life in Tension-Type Headache
Acronym: MTheadacheQL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, PhD, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: ID004
Record Dates: First submitted 2015-03-20; First posted 2015-05-27 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Quality of Life
Keywords: Efficacy; Tension-type headache; Manual therapy
MeSH Terms: conditions — Tension-Type Headache | interventions — Combined Modality Therapy; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Suboccipital inhibitory (Experimental): Suboccipital inhibitory pressure technique. According to this technique, the suboccipital musculature is palpated until contact is made with the posterior arch of the atlas, and progressive and deep gliding pressure is applied, pushing the atlas anteriorly. The occiput rests on the hands while the atlas is supported by the fingertips. Finger pressure must be maintained for 10 minutes to produce the therapeutic effect of inhibiting the suboccipital soft tissues.
  Interventions: Other: Suboccipital inhibitory
- Spinal Manipulative (Experimental): Suboccipital inhibitory pressure technique. This technique is performed along an imaginary vertical line passing through the odontoid process of the axis. No flexion or extension and very little lateroflexion are used. Application is bilateral. First, cephalic decompression is performed lightly, followed by small circumductions. Selective tension is applied to take up tissue slack and create a firm joint barrier. Manipulation is then performed with rotation towards the manipulated side in a helicoidal cranial movement. This technique is designed to correct a generalized dysfunction with the aim of restoring occiput, atlas, and axis joint mobility.
  Interventions: Other: Spinal manipulative
- Combined treatment (Experimental): Consisted in applying the above two techniques using exactly the same sequence: first the SI technique, and then the SM technique.
  Interventions: Other: Combined treatment
- Control group (Placebo Comparator): The subjects received no treatment, but attended the same number of sessions, maintaining the resting position for longer than the experimental groups, and underwent the same evaluations (test for arterial compromise, and the three assessments).
  Interventions: Other: Control group.

INTERVENTIONS:
Other: Suboccipital inhibitory — According to this technique, the suboccipital musculature is palpated until contact is made with the posterior arch of the atlas, and progressive and deep gliding pressure is applied, pushing the atlas anteriorly. The occiput rests on the hands while the atlas is supported by the fingertips. Finger pressure must be maintained for 10 minutes to produce the therapeutic effect of inhibiting the suboccipital soft tissues. The aim is to suppress spasm of the muscles and in general of the suboccipital soft tissues which are responsible for any dysfunctional mobility of the occiput, atlas, or even the axis.
  Arms: Suboccipital inhibitory
Other: Spinal manipulative — This technique is performed along an imaginary vertical line passing through the odontoid process of the axis. No flexion or extension and very little lateroflexion are used. Application is bilateral. First, cephalic decompression is performed lightly, followed by small circumductions. Selective tension is applied to take up tissue slack and create a firm joint barrier. Manipulation is then performed with rotation towards the manipulated side in a helicoidal cranial movement. This technique is designed to correct a generalized dysfunction with the aim of restoring occiput, atlas, and axis joint mobility
  Arms: Spinal Manipulative
Other: Combined treatment — Consisted in applying the above two techniques using exactly the same sequence: first the SI technique, and then the SM technique.
  Arms: Combined treatment
Other: Control group. — The subjects received no treatment, but attended the same number of sessions, maintaining the resting position for longer than the experimental groups, and underwent the same evaluations (test for arterial compromise, and the three assessments).
  Arms: Control group

SUMMARY:
The present study aims to assess the quality of life of patients suffering from tension-type headache (TTH) treated for 4 weeks with different manual therapy-based techniques. The study design involved a factorial, randomized, double-blind, controlled study

DETAILED DESCRIPTION:
Object: The present study aims to assess the quality of life of patients suffering from tension-type headache (TTH) treated for 4 weeks with different manual therapy-based techniques.

Methods: The study design involved a factorial, randomized, double-blind, controlled study of 76 subjects. They were divided into 4 groups: suboccipital inhibitory pressure was applied to the first group; suboccipital spinal manipulation was applied to the second group; a combination of the two treatments was applied to the third group; and the fourth group was a control group. Quality of life was assessed using the SF-12 questionnaire (both overall and in its different dimensions) at the beginning and at the end of treatment, and after one month as a follow-up.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed by a neurologist, with headache characteristics as established by the International Headache Society and Controlled pharmacologically.

Exclusion Criteria:

* Patients with infrequent ETTH, or with probable frequent and infrequent forms of TTH They can never have vomiting or headache episodes during the treatment ETTH patients may experience very occasionally photophobia or phonophobia during their episodes of headache, CTTH patients may experience very occasionally photophobia, phonophobia or mild nausea during headache episodes. Pain aggravated by movement of the head, Metabolic or musculoskeletal problems with similar headache symptoms, Previous trauma to the cervical spine, Active vertigo history Poorly controlled hypertension, Joint stiffness, atherosclerosis, or advanced osteoarthritis, Patients undergoing pharmacological adaptation, Excessive emotional stress, Patients with heart devices Joint instability, Neurological disorders, Laxity of cervical soft tissues, Radiographic abnormalities Generalized hyperlaxity or hypermobility, Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-03; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
frequency of pain | one month prior to the study
  These included major aspects for TTH verification, including frequency of noted pain (less than 15 days monthly = ETTH; more than 15 days monthly = CTTH) response to the classification of the IHS.
severity of pain | one month prior to the study
  These included major aspects for TTH verification, including severity of pain response to the classification of the IHS.

SECONDARY OUTCOMES:
quality of life | 8 weeks
  To assess the subject's quality of life, we applied the health status questionnaire SF-12v2 (Short Form 12 Health Survey) which has shown to be highly reliable. This questionnaire has been adapted to the Spanish context by Alonso et al. and Monteagudo et al.

CONTACTS AND LOCATIONS:
Overall Officials: Gemma V Espí-López, PhD, Study Director — Department of Physiotherapy
Locations (1):
- Gemma v. Espí López, Valencia, Valencia, Spain

REFERENCES:
- [Background] Couppe C, Torelli P, Fuglsang-Frederiksen A, Andersen KV, Jensen R. Myofascial trigger points are very prevalent in patients with chronic tension-type headache: a double-blinded controlled study. Clin J Pain. 2007 Jan;23(1):23-7. doi: 10.1097/01.ajp.0000210946.34676.7d. PMID 17277641
- [Background] Toro-Velasco C, Arroyo-Morales M, Fernandez-de-Las-Penas C, Cleland JA, Barrero-Hernandez FJ. Short-term effects of manual therapy on heart rate variability, mood state, and pressure pain sensitivity in patients with chronic tension-type headache: a pilot study. J Manipulative Physiol Ther. 2009 Sep;32(7):527-35. doi: 10.1016/j.jmpt.2009.08.011. PMID 19748404
- [Background] Espi-Lopez GV, Rodriguez-Blanco C, Oliva-Pascual-Vaca A, Benitez-Martinez JC, Lluch E, Falla D. Effect of manual therapy techniques on headache disability in patients with tension-type headache. Randomized controlled trial. Eur J Phys Rehabil Med. 2014 Dec;50(6):641-7. Epub 2014 Apr 30. PMID 24785463